CLINICAL TRIAL: NCT04373148
Title: Understanding Immunity to SARS-CoV-2, the Coronavirus Causing COVID-19
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Cancer Institute (NCI) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Kari Christine Nadeau, MD, PhD, Professor of Medicine, Stanford University
Other Study IDs: IRB-55689; 2U19AI057229 (NIH); 1U54CA260517-01 (NIH); 1R21ES033049-01 (NIH)
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Coronavirus
Keywords: Immunity
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample and optional nasopharyngeal swab, cheek swab with saliva collection, nasal swab, stool sample, blood microsample, and endotracheal aspirate (sputum samples)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: Participants diagnosed with COVID-19
  Interventions: Other: There is no intervention
- Controls: Participants not diagnosed with COVID-19
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
The purpose of this study is to test over time immunity to SARS-CoV-2, a recently identified coronavirus responsible for the 2019 world-wide pneumonia outbreak known as COVID-19. Adults and children diagnosed with COVID-19 as well as controls without COVID-19 will be invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older) and children with confirmed COVID-19 (RT-PCR diagnosis).
* Adults (18 years and older) and children without COVID-19 for controls (who test negative for COVID-19 but may have viral symptoms)

Exclusion Criteria:

* Patients with special risks attendant to venipuncture will be excluded.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults (18 years and older) and children diagnosed and not diagnosed (controls) with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Testing Immunity to SARS-CoV-2 over time | 1 year

SECONDARY OUTCOMES:
Testing the virus over time | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kari Nadeau, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford Health Care - ValleyCare, Pleasanton, California
  - Stanford University, Hospital, and Clinics, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jia X, Cao S, Lee AS, Manohar M, Sindher SB, Ahuja N, Artandi M, Blish CA, Blomkalns AL, Chang I, Collins WJ, Desai M, Din HN, Do E, Fernandes A, Geng LN, Rosenberg-Hasson Y, Mahoney MR, Glascock AL, Chan LY, Fong SY; CLIAHUB Consortium; Chan Zuckerberg Biohub; Phelps M, Raeber O; Stanford COVID-19 Biobank Study Group; Purington N, Roltgen K, Rogers AJ, Snow T, Wang TT, Solis D, Vaughan L, Verghese M, Maecker H, Wittman R, Puri R, Kistler A, Yang S, Boyd SD, Pinsky BA, Chinthrajah S, Nadeau KC. Anti-nucleocapsid antibody levels and pulmonary comorbid conditions are linked to post-COVID-19 syndrome. JCI Insight. 2022 Jul 8;7(13):e156713. doi: 10.1172/jci.insight.156713. PMID 35801588